CLINICAL TRIAL: NCT00120549
Title: Prospective Randomized Trial of Assisted Hatching of Cleavage Stage Embryos
Brief Title: Study of Assisted Hatching of Cleavage Stage Embryos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shady Grove Fertility Reproductive Science Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1588 WIRB
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2005-07-19 (Estimated); Status verified 2005-07

CONDITIONS: Infertility
Keywords: Assisted Hatching; Cleavage Stage, Ovum; Embryo Transfer; Pregnancy; Embryo Implantation
MeSH Terms: conditions — Infertility

INTERVENTIONS:
Procedure: Assisted embryo hatching

SUMMARY:
The purpose of this study was to determine if assisted embryo hatching can improve pregnancy rates for good prognosis patients undergoing in vitro fertilization (IVF) with day 3 embryo transfer.

DETAILED DESCRIPTION:
Assisted hatching is a procedure in which a hole is made in the hard covering of a developing embryo to allow the embryo to hatch more easily from this shell. This procedure is sometimes used before transferring embryos to patients after in vitro fertilization (IVF) in an attempt to improve resulting pregnancy rates. Assisted hatching has been shown to improve outcomes among certain groups of patients, such as older patients or patients with a history of IVF treatment and embryo transfer without success. Whether this procedure could benefit the broader patient population remains unclear. The purpose of this study was to evaluate potential benefits of assisted hatching for good prognosis patients who would not typically be treated with assisted hatching under current standard protocols. Pregnancy rates were compared between good prognosis patients undergoing IVF with day-3 embryo transfer with or without assisted hatching of the transferred embryos.

ELIGIBILITY:
Inclusion Criteria:

* IVF patients with day 3 embryo transfer
* Maximum age of 39 years
* Maximum FSH 9 mIU/ml
* Maximum E2 75 pg/ml
* Ovulatory menstrual cycles
* Good embryo quality

Exclusion Criteria:

* Diagnosis of diminished ovarian reserve, polycystic ovarian syndrome, uterine or egg factor infertility
* More than one previous unsuccessful IVF cycle

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 2001-08; Study Completion 2005-03

PRIMARY OUTCOMES:
Clinical pregnancy (with fetal cardiac activity) at 5 to 6 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Widra, MD, Principal Investigator — Shady Grove Fertility Reproductive Science Center
Locations (1):
- Shady Grove Fertility Reproductive Science Center, Rockville, Maryland, United States